CLINICAL TRIAL: NCT01972724
Title: A 24-Week, Open Label, Phase IV Trial to Evaluate the Efficacy of Pioglitazone 30 mg in Patients With Inadequately Controlled Type 2 Diabetes Mellitus Treated With Stable Triple Oral Therapy of Metformin, Sulfonylurea, and Pioglitazone 15 Mg (ADD Trial)
Brief Title: Efficacy of Pioglitazone in Participants With Inadequately Controlled Type 2 Diabetes Mellitus Treated With Stable Triple Oral Therapy
Acronym: ADD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG-9999-301-KR; U1111-1145-8222 (Other: World Health Organization)
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-08

CONDITIONS: Type II Diabetes Mellitus
Keywords: Drug therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pioglitazone 15 mg (Double-Blind) (Experimental): Pioglitazone 15 mg tablets, orally, once daily, and metformin and sulfonylurea administered according to the prescribing information of the approved Korean label, for up to 24 weeks.
  Interventions: Drug: Pioglitazone; Drug: Metformin; Drug: Sulfonylurea
- Pioglitazone 30 mg (Double-Blind) (Experimental): Pioglitazone 30 mg tablets, orally, once daily, and metformin and sulfonylurea administered according to the prescribing information of the approved Korean label, for up to 24 weeks.
  Interventions: Drug: Pioglitazone; Drug: Metformin; Drug: Sulfonylurea
- Pioglitazone 30 mg (Open-Label) (Experimental): Pioglitazone 30 mg tablets, orally, once daily, and metformin and sulfonylurea administered according to the prescribing information of the approved Korean label, for up to 24 weeks.
  Interventions: Drug: Pioglitazone; Drug: Metformin; Drug: Sulfonylurea

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone tablets
  Other Names: ACTOS
Drug: Metformin — Metformin as prescribed in clinical practice
Drug: Sulfonylurea — Sulfonylurea as prescribed in clinical practice

SUMMARY:
The purpose of this study is to evaluate the efficacy of pioglitazone 30 mg on glycemic control when used in participants with inadequately controlled type 2 diabetes mellitus treated with stable combinations of metformin and sulfonylurea.

DETAILED DESCRIPTION:
The drug being tested in this study is called pioglitazone. Pioglitazone is being tested to treat glycemic control in adults with inadequately controlled type 2 diabetes mellitus. This study will look at glycemic control in people who take triple oral therapy of metformin, sulfonylurea, and pioglitazone 15 mg.

The study will enroll approximately 114 patients. All participants will be asked to take one pioglitazone tablet at the same time each day throughout the study as well as continuing their previous dose of metformin and sulfonylurea.

This multi-center trial will be conducted in Korea. The overall time to participate in this study is up to 25 weeks. Participants will make 4 visits to the hospital or endocrinologist's office, and will be contacted by telephone 7 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria

Participants meeting the following criteria will be considered for inclusion in the study:

1. Institutional Review Board (IRB)-approved written informed consent form (ICF) must be obtained from the participant or legally authorized representative prior to any trial related procedure (including withdrawal of prohibited medication, if applicable).
2. Participants with a history of clinical diagnosis of established type 2 diabetes mellitus defined by the American Diabetes Association (ADA) criteria 2012.
3. Male or female between 18 and 80 years of age.
4. Participants with stable triple oral therapy of metformin + sulfonylurea + pioglitazone (ACTOS) 15 mg or ACTOSMET(Pioglitazone 15mg/Metformin 850mg) and sulfonylurea for at least 12 weeks at the screening visit.
5. Participants with glycosylated hemoglobin (HbA1c) ≥7.0% at the screening visit.
6. Participants with C-peptide ≥1.0 ng/mL at the screening visit.
7. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from screening throughout the duration of the study, up to 30 days after the last dose of the study medication.

Exclusion Criteria

Participants meeting any of the following criteria will be excluded from enrollment:

1. Participants with type 1 diabetes mellitus or secondary forms of diabetes.
2. Participants who have been treated with insulin for ≥7 days within 3 months prior to the screening visit.
3. Participants with a history of bladder cancer or participants with active bladder cancer.
4. Participants with a history of acute diabetic complications such as diabetic ketoacidosis.
5. Participants with a history of acute or chronic metabolic acidosis, including diabetic ketoacidosis.
6. Participants with unstable or rapidly progressive diabetic retinopathy, nephropathy (estimated glomerular filtration rate [eGFR] <60mL/min/1.73m2).
7. Participants with cardiac insufficiency (e.g., a myocardial infarction, a coronary angioplasty or bypass graft, unstable angina, transient ischemic attacks, or a documented cerebrovascular accident within 6 months prior to the screening visit).
8. Participants with cardiac failure or history of cardiac failure (New York Heart Association [NYHA] Stages 3 to 4).
9. Participants with a serum alanine transaminase (ALT) level ≥2.5 times the upper limit of normal (ULN), active liver disease, or jaundice.
10. Participants taking concomitant gemfibrozil or other strong cytochrome P450 (CYP)2C8 inhibitors.
11. Participants with a history of recurrent or severe hypoglycemia.
12. Participants with a history of any hemoglobinopathy (such as hemolytic anemias or sickle cell disease) that may affect determination of HbA1c.
13. Participants with uninvestigated microscopic hematuria
14. Participants with genetic problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption, since the study drug contains lactose.
15. Participants with any other condition judged by the Investigator as unsuitable for the study.
16. Participants who have used any investigational or experimental drugs or devices within 60 days of the screening visit.
17. Lactating or pregnant female. A positive pregnancy test before the first administration of investigational medicinal product (IMP) or breastfeeding.
18. Male participants planning to father during clinical trial conduct or within 3 months after the last planned dose of the IMP.
19. Participants were previously enrolled into the current clinical trial.
20. The participants participated in the active treatment phase of another clinical trial where a persisting pharmacodynamic effect of the IMP of that clinical trial cannot be excluded.
21. Participants are considered unable or unwilling to co-operate adequately, i.e., to follow clinical trial procedures after Investigator has adequately instructed (e.g., language difficulties, etc.) or participants are anticipated not to be available for scheduled clinical trial visits/procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2016-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (9):
- South Korea (9):
  - Chagwon
  - Daegu
  - Daejeon
  - Gwangju
  - Gyeonggi-do
  - Jeonju
  - Seoul
  - Ulsan
  - Wŏnju

REFERENCES:
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 15 investigative sites in Korea from 16 December 2013 to 17 October 2016.
Pre-assignment Details: Participants with a diagnosis of Type 2 Diabetes Mellitus were enrolled equally in one of 2 treatment groups in the Double-Blind study: pioglitazone15 mg + metformin + sulfonylurea or pioglitazone pioglitazone 30 mg plus metformin + sulfonylurea. Participants received pioglitazone 30 mg + metformin + sulfonylurea in the Open Label study.
Period: Double-Blind
Arm/Group | Pioglitazone 15 mg (Double-Blind) | Pioglitazone 30 mg (Double-Blind) | Pioglitazone 30 mg (Open-Label)
Started | 19 | 18 | 0
Intent-to-treat:Received Study Drug | 17 | 17 | 0
Completed | 10 | 9 | 0
Not Completed | 9 | 9 | 0
Not completed — Rescue Criteria Met | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal of Consent | 2 | 1 | 0
Not completed — Significant Protocol Deviation | 5 | 8 | 0
Period: Open-Label
Arm/Group | Pioglitazone 15 mg (Double-Blind) | Pioglitazone 30 mg (Double-Blind) | Pioglitazone 30 mg (Open-Label)
Started | 0 | 0 | 77
Completed | 0 | 0 | 72
Not Completed | 0 | 0 | 5
Not completed — Withdrew Consent | 0 | 0 | 3
Not completed — Significant Protocol Deviation | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: ITT population included participants who took at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pioglitazone 15 mg (Double-Blind) | Pioglitazone 30 mg (Double-Blind) | Pioglitazone 30 mg (Open-Label) | Total
Number analyzed (Participants) | 17 | 17 | 77 | 111
Age, Continuous [Mean (Full Range); unit: years] | 59.6 (8.73) [44 to 75] | 57.0 (12.0) [31 to 74] | 59.2 (7.88) [39 to 76] | 58.6 [31 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 35 | 51
  Male | 8 | 10 | 42 | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 17 | 17 | 77 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 17 | 17 | 77 | 111
Region of Enrollment [Count of Participants; unit: Participants]
  Korea, Republic Of | 17 | 17 | 77 | 111
Height [Mean (Full Range); unit: cm] | 161.94 (8.392) [147.0 to 175.0] | 163.50 (9.702) [151.0 to 185.0] | 163.25 (9.148) [145.9 to 182.5] | 162.89 [145.9 to 185.0]
Weight [Mean (Full Range); unit: kg] | 70.39 [48.0 to 97.0] | 71.20 [47.5 to 100.0] | 70.38 [46.3 to 101.0] | 70.65 [46.3 to 101.0]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] | 26.86 [22.2 to 36.7] | 26.46 [20.9 to 30.8] | 26.25 [19.0 to 34.6] | 26.52 [19.0 to 36.7]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 24
Description: The change from baseline in glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at Week 24. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population was defined as all participants who took at least 1 dose of the study drug. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Pioglitazone 15 mg (Double-Blind) | Pioglitazone 30 mg (Double-Blind) | Pioglitazone 30 mg (Open-Label)
Number analyzed (Participants) | 17 | 17 | 76
percentage of glycosylated hemoglobin | -0.0003 (0.00725) | -0.0030 (0.00894) | -0.0275 (0.21126)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose at Week 24
Description: The change between the value of fasting serum glucose collected at Week 24 and fasting serum glucose collected at baseline. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 24
Population: Intent-to-treat population was defined as all participants who took at least 1 dose of the study drug.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pioglitazone 15 mg (Double-Blind) | Pioglitazone 30 mg (Double-Blind) | Pioglitazone 30 mg (Open-Label)
Number analyzed (Participants) | 17 | 17 | 77
mmol/L | 0.6727 (1.80662) | -0.4278 (1.88067) | -0.4412 (2.30378)

ADVERSE EVENTS:
Time Frame: First dose of study drug up to 30 days after the last dose of study drug (Up to Week 28)
Description: At each visit investigator had to document any occurrence of adverse events (AEs) and abnormal laboratory findings. Any event spontaneously reported by participant or observed by investigator was recorded, irrespective of relation to study treatment. For other AEs a result of 0 in the table means there are no participants at a threshold of >=5%.
Arm/Group | Pioglitazone 15 mg (Double-Blind) | Pioglitazone 30 mg (Double-Blind) | Pioglitazone 30 mg (Open-Label)
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/17 | 3/77
Other Adverse Events (participants affected / at risk) | 3/17 | 7/17 | 0/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone 15 mg (Double-Blind) (N=17) | Pioglitazone 30 mg (Double-Blind) (N=17) | Pioglitazone 30 mg (Open-Label) (N=77)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pioglitazone 15 mg (Double-Blind) (N=17) | Pioglitazone 30 mg (Double-Blind) (N=17) | Pioglitazone 30 mg (Open-Label) (N=77)
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Oedema (General disorders) | 0 | 2 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0
Onychomycosis (Infections and infestations) | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Venom poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.